CLINICAL TRIAL: NCT01836081
Title: Respirophasic Carotid Artery Peak Velocity Variation as a Predictor of Fluid Responsiveness in Patients With Coronary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2011-0687
Record Dates: First submitted 2013-04-10; First posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Occlusive Disease
Keywords: fluid responsiveness; carotid artery peak velocity variation; coronary disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fluid responsiveness (Experimental)
  Interventions: Other: Volume expansion

INTERVENTIONS:
Other: Volume expansion
  Other Names: volume expansion with 6 mL/kg of 6% hydroxylethyl starch 130/0.4

SUMMARY:
The aim of this study is to investigate usefulness of the respirophasic variation in carotid artery peak flow velocity measured by Doppler ultrasound, which is noninvasive and easily accessible, as a predictor of fluid responsiveness in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. patients scheduled for elective isolated off-pump coronary artery bypass graft surgery

Exclusion Criteria:

1. cardiac rhythm other than sinus
2. congestive heart failure
3. left ventricular ejection fraction <35%
4. history of transient ischemic attack
5. pre-existing cerebrovascular disease and peripheral arterial occlusive disease
6. presence of carotid artery stenosis >50%

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Predictive power of the respirophasic carotid flow peak velocity variation for the fluid responsiveness | Measurement of respirophasic carotid flow peak velocity variation before the volume expansion
  After induction of anesthesia, peak velocity of carotid artery blood flow is measured by the pulsed wave Doppler signal obtained from the left common carotid artery. Respirophasic variation of the peak velocity is defined as the difference between the maximum and the minimum values of peak velocity divided by the mean of the two values during one respiratory cycle. Fluid responder is defined as a patient whose stroke volume index is increased ≥15% after volume expansion. The receiver operating characteristic curve analysis to descriminiate fluid responder is performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Song Y, Kwak YL, Song JW, Kim YJ, Shim JK. Respirophasic carotid artery peak velocity variation as a predictor of fluid responsiveness in mechanically ventilated patients with coronary artery disease. Br J Anaesth. 2014 Jul;113(1):61-6. doi: 10.1093/bja/aeu057. Epub 2014 Apr 9. PMID 24722322